CLINICAL TRIAL: NCT02147886
Title: A Single-Center, Randomized, Double-Blind, Parallel-Group, Dose-Controlled Study, to Assess Safety, Tolerability and Efficacy of Intravenous Cabaletta® in Patients With Machado-Joseph Disease
Brief Title: Study To Assess Safety, Tolerability and Efficacy of Intravenous Cabaletta in Patients With Machado-Joseph Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bioblast Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BB-MJD-201
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Machado-Joseph Disease / Spinocerebellar Ataxia 3
Keywords: Bioblast, Randomized, parallel-group, and dose-controlled
MeSH Terms: conditions — Machado-Joseph Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cabaletta 15gr (Experimental): Cabaletta 15gr
  Interventions: Drug: Cabaletta for IV infusion once weekly during 24 weeks
- Cabaletta 30gr (Experimental): Cabaletta 30gr
  Interventions: Drug: Cabaletta for IV infusion once weekly during 24 weeks

INTERVENTIONS:
Drug: Cabaletta for IV infusion once weekly during 24 weeks — Cabaletta for IV infusion once weekly
  Arms: Cabaletta 15gr
Drug: Cabaletta for IV infusion once weekly during 24 weeks
  Arms: Cabaletta 30gr

SUMMARY:
* This is an exploratory, randomized, parallel-group, dose escalation and dose-controlled study without a placebo arm.
* Eligible patients will be randomized in a 1:1 ratio (double-blind) to receive Cabaletta in 2 doses, once weekly for 22 weeks (total of 24 weeks of treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, 18 - 75 years
2. Clinically diagnosed as Machado-Joseph disease/Spinocerebellar ataxia 3 confirmed by genetic testing
3. With disease stage 2 or less
4. Stable doses of all medications for 30 days prior to study entry and for the duration of the study.
5. Body Mass Index (BMI) ≤32 kg/m2.
6. Ability to ambulate with or without assistance

Exclusion Criteria:

1. Diabetes mellitus type 1 or 2
2. Other major diseases
3. Uncontrolled heart disease, chronic heart failure (CHF).
4. Other neurological diseases.
5. Ataxia derived from any other cause than genetically-confirmed spinocerebellar ataxia
6. Presence of psychosis, bipolar disorder, untreated depression
7. History of malignancy (except non-invasive skin malignancy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Adverse events | 28 weeks
  Safety will be evaluated on the basis of the following assessments:
  Adverse events , physical examination, 12-lead ECG, vital signs, safety laboratory evaluations
Physical examination | 28 weeks
  Safety will be evaluated on the basis of the following assessments:
  Adverse events , physical examination, 12-lead ECG, vital signs, safety laboratory evaluations
Vital signs | 28weeks
  Safety will be evaluated on the basis of the following assessments:
  Adverse events , physical examination, 12-lead ECG, vital signs, safety laboratory evaluations
12-lead ECG | 28weeks
  Safety will be evaluated on the basis of the following assessments:
  Adverse events , physical examination, 12-lead ECG, vital signs, safety laboratory evaluations
Safety laboratory tests | 28weeks
  Safety will be evaluated on the basis of the following assessments:
  Adverse events , physical examination, 12-lead ECG, vital signs, safety laboratory evaluations

SECONDARY OUTCOMES:
Disease markers | 27 weeks
  Changes in disease markers will be assessed based on the following assessments:
  Scale for the Assessment and Rating of Ataxia (SARA); Neurological Examination Score for Spinocerebellar Ataxia (NESSCA); Change in BMI - screening, spinocerebellar Ataxia Functional Tests; quality of life

OTHER OUTCOMES:
Biochemical marker | 27 weeks
  Assessment of disease biochemical marker neuron specific enolase (NSE) and protein S 100 B (S100B)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gordon, Prof., Principal Investigator — Meir Medical Center Kfar Saba Israel
Locations (1):
- Meir Medical Center, Kfar Saba, Israel